CLINICAL TRIAL: NCT06886191
Title: Effects on Urine Oxygenation of Forced Diuresis with Neutral Fluid Balance During Cardiac Surgery, a Randomized Controlled Trial
Brief Title: PuO2 in RenalGuard Pilot Study
Acronym: PURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahlgrenska University Hospital (Other)
Responsible Party: Principal Investigator, Lukas Lannemyr, Consultant Anesthesiologist, MD, PhD, Sahlgrenska University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PUREstudy
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Cardiac Surgery Subjects
Keywords: renal oxygenation; urine oxygen tension; furosemide; balanced diuresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- RenalGuard (RG) (Experimental): The RG system is used to ensure neutral (0) fluid balance while maintaining a urine flow >200 ml/hour. Urine output is replaced 1:1 with Plasmolyte solution. In patients randomized to RG, therapy is initiated after baseline measurements but before the start of surgery.
  If baseline urine flow is < 200 ml/hour, a bolus dose of furosemide (20 mg iv) is given, and additional furosemide bolus and/or titration of continuous furosemide infusion may be given to maintain urine flow rate >200ml/hour.
  After completed surgery, RG therapy continues until 3 hours after weaning from CPB
  Interventions: Device: RenalGuard Therapy
- Standard of Care (No Intervention): Conduct of cardiopulmonary bypass will be done according to local clinical practice

INTERVENTIONS:
Device: RenalGuard Therapy — Fluid management system, which weighs urine and controls intravenous administration of crystalloid solution.
  Arms: RenalGuard (RG)

SUMMARY:
The PuO2 in RenalGuard (PURE) study is planned as a single center, randomized controlled pilot study comparing renal oxygenation during cardiac surgery with cardiopulmonary bypass (CPB) with or without balanced forced diuresis using the RenalGuard (RG) system.

Renal oxygenation will be assessed by urine oxygen tension, continuously measured by optodes placed through the urine catheter. Measurements will start after induction of anesthesia and continue for 24 hours.

In total, 30 patients will be randomized 1:1 to RG or standard of care (SOC) during cardiac surgery with CPB. In the RG group, the forced diuresis with neutral fluid balance will be maintained from before the start of surgery until 3 hours after weaning from CPB.

The primary endpoint is the group difference (RG vs SOC) in delta PuO2, defined as the change in mean PuO2 from baseline to the last 5-minute period at 45 minutes after start of CPB.

The secondary endpoints include

1. Group difference in mean PuO2 before, during and after CPB
2. Group difference in time weighted area under the curve for PuO2
3. Group differences in renal near infrared spectroscopy (NIRS) before, during and after CPB
4. Group difference in urine and blood biochemistry including renal biomarkers
5. Group difference in urine output and fluid balance during surgery and first postoperative day
6. Group differences in postoperative AKI according to the KDIGO criteria
7. Time (minutes) with puO2 ≤ 15 and ≤ 10 mmHg during and after CPB
8. Dynamics of PuO2 during the early postoperative phase

Patients ≥18 years scheduled for cardiac surgery with CPB with estimated glomerular filtration rate ≥50 ml/min are eligible for inclusion. Exclusion criteria include patients on higher doses of furosemide, patients with AKI or under renal replacement therapy.

Patients will be analyzed according to study group. In patients where hemofiltration has been used during CPB, control group patients who has received furosemide and patients in the RG group who do not reach target urine flow will be excluded from the main analysis but will be included in a separate analysis.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥18 years of age
* scheduled for cardiac surgery with normothermic CPB
* Estimated glomerular filtration rate ≥50 ml/min as assessed by the CKD-EPI formula

Exclusion Criteria:

* Patient receiving furosemide at a dose>100 mg/day orally (or the equivalent dose of an alternative loop diuretic) in the last week
* Patient who cannot be urethrally catheterized for any reason
* Patient already dialysis dependent
* Known or suspected AKI (KDIGO criteria) at the time of screening
* Any condition which, in the judgement of the investigator, might increase the risk to the patient

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-03-17 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Delta PuO2 | Baseline (before start of surgery) to 45 minutes after start of CPB
  The primary endpoint is the group difference (RG vs controls) in delta PuO2, defined as the change in mean PuO2 from baseline to the last 5-minute period at 45 minutes after start of cardiopulmonary bypass (CPB) (or the last 5 minutes if cross clamp release is done before)

SECONDARY OUTCOMES:
Repeated PuO2 | baseline, 30, 45 minutes on CPB and at 30, 60 and 240 minutes after CPB
  Group difference in mean PuO2 at specified times
PuO2 AUC | From baseline before start of surgery until 4 hours after CPB
  Group difference in time weighted area under the curve (AUC) for PuO2 during CPB and until removal of the PuO2 measurement
PuO2 sub threshold | From baseline before surgery until 4 hours after CPB
  Time (minutes) with puO2 ≤ 15 and ≤ 10 mmHg during and after CPB
Diuresis and fluid balance | 24 hours
  Diuresis and net fluid balance (incorporating fluids given and lost) during surgery and during the first 24 hours.

OTHER OUTCOMES:
Dynamics of PuO2 during the early postoperative phase | 24 hours
  Repeated measurements of PuO2 during the first postoperative 24 hours.
Urine Nephrocheck | 4 hours after CPB
  Urine IGFBP2*TIMP2 at 4 hours after Cardiac surgery
Renal near-infrared spectroscopy (NIRS) | From baseline before surgery until 4 hours after CPB
  Group differences in renal NIRS at baseline, 30 minutes on CPB and at 30, 60 and 240 minutes after CPB
Creatinine | 7 days
  Development of serum creatinine from baseline and daily for up to seven postoperative days

CONTACTS AND LOCATIONS:
Overall Officials: Lukas Lannemyr Lannemyr, MD, PhD, Principal Investigator — Institute of Clinical Sciences, Dept of Anesthesia and Intensive Care, Sahlgrenska Academy, Gothenburg University. Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: Undecided
Parts of the data may be analyzed in other projects